CLINICAL TRIAL: NCT05077150
Title: A Case-control Study on Risk Factors, Timing, and PCR Use, for Pneumocystis Pneumonia (PcP) After Allogeneic HSCT
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: (4)8414112
Record Dates: First submitted 2017-01-06; First posted 2021-10-14 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Pneumocystis Pneumonia
Keywords: jirovecii; pneumocystis; PCP
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCP cases: Any allogeneic HSCT recipient who, during the 1-year study period, underwent a BAL from the day of transplant, and whose BAL fluid was positive for PcP: either by qPCR alone, or positive cytology or IF, irrespectively of clinical presentation, imaging, co-infection and PcP treatment. Only first episode of PcP will be included (incident cases).
  Due to the lack of standardization, qPCR on sputum only will not be taken in account for the diagnosis of PcP.
- Controls: Controls are matched to case on Centre and HSCT date and if possible on gender and date of birth.

SUMMARY:
The fungus Pneumocystis jirovecii is responsible for pneumocystosis (PcP), a life threatening pneumonia in patients undergoing HSCT. The spontaneous attack rate of 16% within the first 6 months following allogeneic HSCT reported in the 1980's has considerably decreased with prophylaxis. However, PcP still remains a concern in the transplant ward with an incidence rate up to 2.5% in allo- and 1.4% in autologous HSCT but up to 7.2% on low dose of Dapsone. The mortality of PcP is especially high in HSCT recipients. One of the main factors of PcP after HSCT seems to be either the lack of TMP-SMX prophylaxis (all the other prophylactic drugs being inferior to TMP-SMX), or poor compliance to prophylaxis. Due to the rarity of the disease after HSCT, it is impossible to study it in monocenter studies, except on very long periods of time which may not reflect current practice. Several questions deserve investigations in a multicenter study, about timing, risk factors, and outcome.

Moreover, some European laboratories involved in the diagnosis of PcP have already given up to classical diagnostic methods and switched to qPCR. This implies that lower fungal burden can be detected and the clinical pertinence of such a diagnostic strategy deserves to be assessed.

DETAILED DESCRIPTION:
Due to the lack of standardization, qPCR on sputum only will not be taken in account for the diagnosis of PcP. Knowing this is a non-interventional study, no additional visits or laboratory tests will be performed for the study. Only the available data will be collected.

ELIGIBILITY:
Inclusion Criteria PCP cases:

* Allogeneic HSCT within the previous 24 months
* New case (first onset) of PcP documented in a BAL fluid, whatever the positive diagnostic test (cytology or IF or PCR) and whatever the presentation and treatment
* Any age
* Pre or post-transplant signed informed consent to enter the data in the EBMT registry

Exclusion Criteria PCP cases:

* Autologous HSCT
* Allogeneic HSCT recipient transplanted more than 24 months at time of the onset of PcP
* Second episode of PcP since allogeneic HSCT (patients who had experienced PcP before the allogeneic HSCT are not excluded).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have received an allogeneic HSCT during the last 24 months and who have a BAL fluid positive for Pneumocystis jirovecii (qPCR or IF or cytology) during the study period will be included, irrespectively of age, transplant characteristics and irrespectively to the fact that the patient has been treated for PcP or not.
  Assuming an incidence of 3% after allogeneic HSCT, a total number of 3 300 allogeneic transplant (roughly 100 centers) would allow to expect 100 cases of PcP.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Post-transplant risk factors for PCP infection | 90 days
  To identify pre- and post-transplant factors associated with development of PcP after allogeneic HSCT including:
  Underlying disease, graft versus host disease, relapse of underlying disease, immune status, co-infections, age

CONTACTS AND LOCATIONS:
Overall Officials: Christine Robin, MD, Principal Investigator — Hematology Department, Pr Cordonnier. henri Mondor University Hospital; Simone Cesaro, MD, Study Chair — Paediatric Haematology Oncology. Policlinico G.B. Rossi
Locations (9):
- University Hospital Gasthuisberg, Leuven, Belgium
- France (4):
  - University of Amiens: CHU Amiens, Amiens
  - Hôpital Henri Mondor, Créteil
  - Hôpital Huriez, Lille
  - Hopital St. Louis, Paris
- University Hospital Eppendorf, Hamburg, Germany
- United St. Istvan and St. Laszlo Hospital, Budapest, Hungary
- Rambam Medical Center, Haifa, Israel
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided